CLINICAL TRIAL: NCT00497900
Title: The Effect of Calcium and Vitamin D in Patients With Heart Failure
Acronym: KarViDII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Louise Lind Schierbeck, MD, research fellow, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-005767-26
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2012-03

CONDITIONS: Heart Failure; Vitamin D Deficiency
MeSH Terms: conditions — Heart Failure; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Calcium and vitamin D
  Interventions: Drug: Vitamin D
- 2 (Placebo Comparator): Calcium and placebo (cellulose)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Daily vitamin D (cholecalciferol) tablets and rocaltrol

SUMMARY:
Previous studies have shown high proportions of vitamin D deficiency among elderly in Denmark. Vitamin D is important for muscular function. The investigators intend to examine if it is possible to improve cardiovascular function in patients with heart failure and vitamin D deficiency by supplementation with vitamin D.

DETAILED DESCRIPTION:
Heart failure (HF) is a major course of morbidity and mortality. The prevalence in the Danish population is 1-2% and for age 50 -75 years: 2-3% (1) . It has been estimated that there are currently 6.5 million HF patients in Europe and 5 million in the USA (2) . Lack of vitamin D has been linked to heart disease including ischemic heart disease, heart failure, and hypertension.(3) Vitamin D deficiency is prevalent in the elderly population. Calcium absorption, bone mineralization and muscle function may be impaired. Vitamin D receptors have also been demonstrated in skeletal as well as cardiac muscle(4) . Vitamin D and Parathyroid Hormone (PTH) are closely linked in the calcium metabolic system. In order to maintain serum calcium within range PTH and vitamin D acts together in response to changes in serum-calcium levels. 25(OH)D concentration also being an important factor determining the levels of PTH.(5) Decreasing vitamin D leads to increasing levels of PTH. Hyperparathyroidism in patients with kidney-disease has in numerous studies been linked to cardiovascular disease, left ventricle hypertrophy, and valvular calcification .(6) Aim: Intervention with vitamin D and calcium will improve patients' vitamin D levels and suppress PTH. Thus we hope to find an improved cardiac function and quality of life in the intervention-group.

Comparison: Cardiac function (and other effect parameters - such as self-evaluated health) in the intervention group vs. in the placebo-group

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Vitamin D (serum 25-OHD): 50nmol/l or less
* Heart failure (EF 40% or less, NYHA:2 or more)

Exclusion Criteria:

* Calcium metabolic disturbances
* Granulomatous diseases
* Alcohol or drug abuse
* Intake of 400IU (or more) vitamin D/day
* Condition too poor to participate
* Pregnancy
* AF with HF 90 or above
* Mitral insufficiency, degree 3 or above
* Large cardiac aneurisms
* Significant aorta stenosis
* Significant aorta insufficiency
* Allergy to components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-08; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | 6 months

SECONDARY OUTCOMES:
6 minutes walk test | 6 months
  combined skeletal and cardiac muscle function
Quality of life | 6 months
  Self assessed health (MLHFQ)
Biochemical markers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Erik B Jensen, MD, PhD, Study Director — Hvidovre University Hospital; Louise Lind Schierbeck, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Background] Nielsen OW, Raymond IE, Kirk V, Pedersen F, Bay-Nielsen M. [The epidemiology of heart failure from a Danish perspective]. Ugeskr Laeger. 2004 Jan 19;166(4):243-7. No abstract available. Danish. PMID 14964101
- [Background] Holick MF. The vitamin D epidemic and its health consequences. J Nutr. 2005 Nov;135(11):2739S-48S. doi: 10.1093/jn/135.11.2739S. PMID 16251641
- [Background] O'Connell TD, Simpson RU. Immunochemical identification of the 1,25-dihydroxyvitamin D3 receptor protein in human heart. Cell Biol Int. 1996 Sep;20(9):621-4. doi: 10.1006/cbir.1996.0081. PMID 8948124
- [Background] Pepe J, Romagnoli E, Nofroni I, Pacitti MT, De Geronimo S, Letizia C, Tonnarini G, Scarpiello A, D'Erasmo E, Minisola S. Vitamin D status as the major factor determining the circulating levels of parathyroid hormone: a study in normal subjects. Osteoporos Int. 2005 Jul;16(7):805-12. doi: 10.1007/s00198-004-1757-4. Epub 2004 Nov 16. PMID 15551058
- [Background] Horl WH. The clinical consequences of secondary hyperparathyroidism: focus on clinical outcomes. Nephrol Dial Transplant. 2004 Aug;19 Suppl 5:V2-8. doi: 10.1093/ndt/gfh1049. PMID 15284353